CLINICAL TRIAL: NCT04342845
Title: Effectiveness of Motivational Interviewing on Improving Care for Patients With Type 2 Diabetes in China: A Randomized Controlled Trial
Brief Title: Effectiveness of Motivational Interviewing on Improving Care for Patients With Type 2 Diabetes in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JCYJ20150331142757385
Record Dates: First submitted 2020-03-30; First posted 2020-04-13 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Motivational interviewing; Patient empowerment; Self-management; China
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Patient Participation

STUDY DESIGN:
Intervention Model Description: Two hundred and twenty-five patients, recruited from community health centers (CHCs) and the family medicine clinic in the University of Hong Kong-Shenzhen Hospital in Shenzhen, were randomly assigned to the intervention or control groups. Patients in the intervention group (n = 117) received a four-session PEP in small groups over 1 month by trained nurses and doctors. The control group (n = 108) received the traditional lecture-style health education on DM. All the patients were followed up for 3 months. Outcomes included problem areas in diabetes (PAID) that measures diabetes-related emotional distress, patient enablement index (PEI), mental health, patient satisfaction respectively as well as lifestyle behaviors were assessed at baseline, post-activity and 3 months.
Who Masked: Participant
Masking Description: Upon receiving a participant's consent form, the independent administrative research assistant would generate a random number by computer to determine allocation to the intervention or control group. For concealment purposes, there was no medical information relating to the participant on the consent form. The assistant only informed participants of their attendance time and not of their grouping. We used the blocked randomization by number "8" which guaranteed that there were four people in both groups in each of the eight people. This method can avoid overbalance between two groups as there might be some people missing halfway.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational interviewing (Experimental): The intervention group received an education program in small groups that included no more than ten members. The content was designed based on MI theory and the theory of patient empowerment. Program content was further informed by the Hospital Authority Patient Empowerment Program in Hong Kong. The education program consisted of four modules, held once a week, that each lasted approximately 1½ to 2 hours. They were grouped under the following four broad headings: Knowing Diabetes, Diabetes Self-Care, Healthy Diet and Physical Exercise. Each module started with a brief introduction to relevant background knowledge, which was followed by small-group discussions about personal barriers and techniques for overcoming challenges. During the small group discussions, educators acted as MI facilitators, using group MI techniques to strengthen participants' motivation.
  Interventions: Behavioral: Experimental: Motivational interviewing Placebo Comparator: Traditional lectures
- Traditional lectures (Placebo Comparator): The control group received traditional lectures that consisted solely of conveying healthcare information to patients. In order to minimize intervention bias, the control group lectures were standardized and adapted into four modules, namely knowing diabetes, healthy diet, physical exercises, and how to use medication correctly, which were similar topic headings, durations and frequencies to those of the intervention group. Each lecture was 1 hour and was provided by one of four health professionals (a pharmacist, dietician, endocrinologist or nurse) who had never received any prior training in MI.
  Interventions: Behavioral: Experimental: Motivational interviewing Placebo Comparator: Traditional lectures

INTERVENTIONS:
Behavioral: Experimental: Motivational interviewing Placebo Comparator: Traditional lectures — Patients in the intervention group (n=117) received a four-session patient empowerment program in small groups over one month by trained nurses and doctors. he control group received traditional lectures that consisted solely of conveying healthcare information to patients.

SUMMARY:
n 2015, the International Diabetes Federation estimated that there were nearly 110 million diabetes mellitus (DM) patients in China, which was the highest number recorded in the world. China's DM-related costs, ranked second highest globally, were estimated to be US$51 billion. In response to the rising patient numbers and costs, the Chinese government has invested heavily in primary healthcare since 2009, with the goal of improving chronic disease management in the primary care settings. A key part of the primary care improvement program prioritizes health education as a route to lifestyle modification. Although the content and modes of delivery vary enormously, most of the programs focused on providing information rather than facilitating patient change. The impacts of traditional patient education on lifestyle modification and changes in psychological status have been reported to be suboptimal. These may be related to the poor understanding of the educational content or lack of means for making changes as a result of low socioeconomic status and poor educational level. It is therefore necessary to rethink and explore a more structured, patient-centered approach to health education at improving the outcomes of DM control.

Motivational interviewing (MI) is a collaborative, patient-centered counseling approach that aims to elicit behavior change. Counselors use empathy and other techniques to create an atmosphere to help patients to explore the discrepancies between the goals and their current behavior. The focus of MI is to find and resolve the ambivalence, improve patients' perception of the importance of behavior change, and support them to make the change. MI provides a structural framework with guiding principles that can be easily followed by the primary care doctors. Some studies show that MI can contribute to improve healthy eating, weight control and increases in physical activity, but most research focused on intermediate outcome measures and did not evaluate the readiness to change. MI can be utilized by a variety of healthcare providers, which makes it adaptable for different culture and clinical settings. However, the effectiveness of MI in Chinese diabetic patients remains uncertain.

MI has been delivered using different methods. These methods have varied and included a single one-to-one session with a therapist, multiple group sessions, and the incorporation of MI into daily clinical practice. Furthermore, in yet another study, MI education program produced a significantly greater change in patients' perceived competence in dealing with diabetes than the control group. In this study, the investigators adopted the group MI approach and developed a patient empowerment program (PEP) utilizing the techniques and framework of MI. The investigators compared this to the most common form of DM education in China, i.e., when health professionals (nurses, doctors, dietitians or pharmacists) give a lecture on DM to patients and their carers in a hospital lecture theatre in a didactic manner.

DETAILED DESCRIPTION:
Background: To assess the effects of a motivational interviewing (MI)-based patient empowerment program (PEP) on type 2 diabetes mellitus (DM) patient self-management compared to traditional diabetes health education.

Methods: Two hundred and twenty-five patients, recruited from community health centers (CHCs) and the family medicine clinic in the University of Hong Kong-Shenzhen Hospital in Shenzhen, were randomly assigned to the intervention or control groups. Patients in the intervention group (n=117) received a four-session PEP in small groups over one month by trained nurses and doctors. The control group (n=108) received the traditional lecture-style health education on DM. All the patients were followed up for three months. Outcomes included problem areas in diabetes (PAID) that measures diabetes-related emotional distress, patient enablement index (PEI), mental health, patient satisfaction respectively as well as lifestyle behaviors were assessed at baseline, post-activity and three months.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with HbA1c between 7-10%, 18-75 years old

Exclusion Criteria:

* Known severe comorbidities or complications, such as cancer, unstable angina, frequent exacerbation of chronic obstructive pulmonary disease, or diabetic retinopathy, Illiterate or not cognitively competent enough to understand written and the oral expression of the language native to the study site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Problem Areas in Diabetes Questionnaire | 4 months
  PAID is a self-administered 20-item scale. Each item is scored from 0 (not a problem) to 4 (serious problem). The PAID scale has been widely used in many countries to assess diabetes-related emotional distress.

SECONDARY OUTCOMES:
"Patient Enablement Index" (PEI) score | 4 months
  The PEI is a scale that measures patients' enablement, it was also used to measure patient enablement in this study. The PEI scale had been validated in the Chinese population.
Stages of Change score | 4 months
  The Stages of Change score is a score that assess participants' readiness to change in behaviors such as smoking, drinking or exercise and their adherence to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jingya Yan, Principal Investigator — WHO Health Promoting Hospital Office, The University of Hong Kong - Shenzhen Hospital, Shenzhen, China.; Wei Liang, Principal Investigator — Endocrinology Department, The University of Hong Kong - Shenzhen Hospital, Shenzhen, China.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF